CLINICAL TRIAL: NCT06336720
Title: Portable Neuromodulation Stimulator (PoNS®) Therapy for Gait and Balance Deficits in Chronic Stroke Survivors: A Single-Arm Study
Brief Title: PoNS® Therapy for Gait and Balance Deficits in Chronic Stroke Survivors: A Single-Arm Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helius Medical Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMI-SA-PoNS-STK001
Record Dates: First submitted 2024-03-18; First posted 2024-03-29 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-09

CONDITIONS: Chronic Stroke Survivors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single Arm (Other): open label administration of translingual neurostimulation.
  Interventions: Device: Portable Neuromodulation Stimulator (PoNS)

INTERVENTIONS:
Device: Portable Neuromodulation Stimulator (PoNS) — The active PoNS device delivers amplitude-controlled, biphasic pulses to the anterior superior surface of the tongue through gold-plated electrodes.

SUMMARY:
Primary Objective: To further evaluate the aspects of safety related to PoNS therapy in chronic stroke survivors.

Secondary Objectives: To further evaluate the efficacy of PoNS on improving dynamic gait and balance, establishing durability of effect, risk of falling and fall rate. As well as adherence to PoNS device utilization.

Exploratory Objectives: To further evaluate quality of life to measure physical, mental, behavioral, and general health, as well as functional decline (> 30% on gait or balance improvement at endpoint) during the 12-week follow-up.

DETAILED DESCRIPTION:
Observational, interventional, single-arm, open label, clinical trial investigating PoNS utilization with combined with dynamic gait and balance rehabilitation exercise (DGB training) in chronic stroke survivors.

6 The data from this prospective, single arm, multi-site, study that will enroll 30 subjects at 3 different clinical sites will be used to augment safety data obtained in the RCT (which will randomize 60 patients 1:1 into either active PoNS combined with DGB training versus DGB training with a sham device). The totality of the proposed clinical evidence spans 3-4 sites and approximately 90 patients.

Eligible study participants in this study will be assigned to treatment with a PoNS device ["active"]. Participants will work with a study physical therapist - trained on PoNS Therapy by HMI Medical and registered as a PoNS Trainer (Trainer). The Trainer will prepare a DGB training exercise program appropriate to the participant's ability level and instruct on how to perform the breathing and awareness (mindfulness) training (BAT). To ensure patient's safety during rehabilitation at home, the Trainer may assign a DGB training program slightly different from the one performed in clinic.

All participants will undergo a total of twelve weeks of DGB training program, performed both in clinic (4 weeks, Part 1), supervised by the Trainer, and at home (8 weeks, Part 2), unsupervised. At the end of the treatment period, they will be asked to return to the clinic site for the follow-up visit 12 weeks after the end of the treatment period, as shown below:

During the training sessions in clinic and, subsequently, during at-home training period, the trainer can adjust /flex the DGB training based on the participant's individual response to PoNS Therapy. During Phase 2, the Trainer will follow-up weekly with participants either in person, or through a telemedicine session, if patient is unavailable to travel to the clinic.

Twelve weeks after completing the 12-week treatment phase of the study, participants will be required to return to the clinic for the final assessment of treatment effect. During the 12-week follow-up period (Part 3), participants will no longer utilize PoNS device but will still be encouraged to continue with their physical rehabilitation program for the duration follow-up period until the final study visit.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 18 and < 85 years of age with a diagnosis ischemic or hemorrhagic stroke at > 6 months since stroke onset event.
2. FMA-LE scores < 34 at screening with residual paresis in the lower extremity.
3. Able to walk at least 10 feet with or without assistive device.
4. FGA score < 23 at screening.
5. Montreal Cognitive Assessment 5-min (MoCA 5-min) ≥ 6
6. Able to understand, learn and apply instructions on how to operate the PoNS device and perform the rehabilitation exercise program.

Exclusion Criteria:

1. Pre-existing neurological disorders or previous stroke affecting the other hemisphere.
2. Severe arthritis or orthopedic problems that limit passive range of motion.
3. Areas of recent bleeding or open wounds; or areas that lack normal sensation on the tongue.
4. Diagnosis of dementia or mild cognitive impairment
5. Concurrent daily use of transcutaneous electric nerve stimulation (TENS) and/or other peripheral stimulation devices (i.e. Bioness®)
6. Neurostimulation therapy over the previous 6 months
7. Cancer treatment within the past year.
8. Nonremovable metal orthodontic devices.
9. Oral health problems.
10. Chronic infectious diseases.
11. Pregnancy.
12. Sensitivity to nickel, gold or copper.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Primary safety endpoints | 12 week
  treatment - related serious adverse events (SAE) over 12 week treatment

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Brooks Rehabilitation, Jacksonville, Florida
  - Shepherd Center, Atlanta, Georgia
  - MGH Institute of Health Professions, Boston, Massachusetts
  - Neurology Center of New England, P.C., Foxborough, Massachusetts
  - Rehabologym Corp, Tarrytown, New York